CLINICAL TRIAL: NCT05121961
Title: Treatment for Sacroiliac Joint Pain Using Platelet-rich Plasma (PRP) Regenerative Therapy: A Randomized Controlled Trial in Comparison With Steroid/Anesthetic Injection With Advanced MR Analysis
Brief Title: Treatment for Sacroiliac Joint Pain Using Platelet-rich Plasma (PRP) Versus Steroid/Anesthetic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Principal Investigator, Miriam Peckham, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSCH1923
Record Dates: First submitted 2021-10-20; First posted 2021-11-16 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain; Sacroiliac Joint Synovitis
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled trial
Who Masked: Participant
Masking Description: Patients will be blinded to which injectate they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-rich Plasma (Experimental): Patients will receive an intra-articular injection 3 mL of autologous platelet-rich plasma in the sacroiliac joint.
  Interventions: Procedure: Sacroiliac intra-articular injection
- Steroid/Anesthetic (Active Comparator): Patients will receive an intra-articular injection 40 mg Depo-medrol mixed with 2 mL 0.25% bupivicaine in the sacroiliac joint.
  Interventions: Procedure: Sacroiliac intra-articular injection

INTERVENTIONS:
Procedure: Sacroiliac intra-articular injection — CT guided injection of platelet-rich plasma versus steroid/anesthetic into the sacroiliac joint

SUMMARY:
The purpose of this study is to determine if platelet-rich plasma is superior to steroid/anesthetic for the treatment of sacroiliac joint pain.

DETAILED DESCRIPTION:
All patients with sacroiliac joint pain diagnosed by a back pain specialist will undergo physical examination maneuvers and a test lidocaine injection of the joint. Patients who meet eligibility requirements will be randomized in a single-blind randomized controlled manner with a 50% chance of receiving platelet-rich plasma versus steroid/anesthetic injection of the sacroiliac joint(s).

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 y/o) males and females referred for therapeutic injection to the investigators spine interventional service by a physiatrist or pain anesthesiologist with a clinical diagnosis of SIJ pain confirmed by history
* 50% or greater reduction in pain by a diagnostic anesthetic block using no more than 1.5 cc 2% lidocaine performed under imaging guidance by a pain interventionalist (PM&R, Pain Anesthesia, or Neuroradiology Spine Intervention).
* Baseline pain must be >/=4 by numeric rating scale (NRS), at least 6 weeks in chronicity, and must not be multi-factorial (related to radiculopathy or axial pain localizing elsewhere) by physical examination or confounding medical history (infection, inflammatory spondyloarthropathy, or osseous metastatic disease).

Exclusion Criteria:

* SIJ steroid treatment within the prior 6 months.
* Patients with a history of infection currently on antibiotic therapy
* Usage of systemic immunosuppressants
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-02-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | Change between baseline and 3-months post-intervention
  Validated pain scale rating pain on a scale of 0 through 10. 0 for no pain, and 10 for the highest pain the patient can imagine.

SECONDARY OUTCOMES:
Modified Oswestry Disability Questionnaire | Change between baseline and 3-months post-intervention
  Validated questionnaire used to evaluate function in patients with low back pain. The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
Short-Form 12 Survey | Change between baseline and 3-months post-intervention
  Validated survey used to evaluate function in patients with low back pain. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Functional testing | Change between baseline and 3-months post-intervention
  2 validated tests for low back pain "get up and go," "5 time sit to stand." Shorter times indicate better physical function, and longer times indicate poorer physical function.
Opiate/pain medication usage questionnaire | Change between baseline and 3-months post-intervention
  Questionnaire on type, dose, and frequency of pain medications being used by the patient. All opiates will be converted to the morphine milligram equivalent scale with lower values indicating lower opiate content and higher values indicating higher opiate content

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Peckham, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - Veterans Administration Salt Lake City Health Care System, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT05121961/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT05121961/ICF_001.pdf